CLINICAL TRIAL: NCT04924972
Title: Face-Q Patient-Report Assisted Subjective and Objective Evaluation of Upper Eye Lid Blepharoplasty Outcomes Using Different Suturing Techniques: A Randomized Observer and Patient-Blinded Pilot Study
Brief Title: FACE-Q in Blepharoplasty
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Told, Clinical Professor, Medical University of Vienna
Other Study IDs: OPHTH-011018
Record Dates: First submitted 2019-08-06; First posted 2021-06-14 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Dermatochalasis of Upper Eyelid
MeSH Terms: interventions — Blepharoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intracutaneous Suture
  Interventions: Procedure: Blepharoplasty
- running Suture
  Interventions: Procedure: Blepharoplasty

INTERVENTIONS:
Procedure: Blepharoplasty — 90 patients undergoing bilateral upper eyelid blepharoplasty are randomly assigned to a suturing technique (running cutaneous or subcuticular Nylon (6-0 Prolene) sutures). Steri-strips will be used until suture removal 7 days after blepharoplasty for patient blinding.

SUMMARY:
The aim of this study is to assess the effect of two different suturing techniques in patients undergoing bilateral upper eyelid blepharoplasty on the results of the FACE-Q Eye Module questionnaire for measuring patient-reported outcomes as well as on the blinded objective assessment by two experienced surgeons using the same questionnaire.

We aim to investigate the differences of the 2 most common techniques of skin closure with running cutaneous or subcuticular Nylon (6-0 Prolene) sutures in upper blepharoplasties and their effect on postoperative complications and scar formation. Besides the functional outcomes (visual field) and objective postoperative results, we aim to measure the patients' satisfaction using the FACE-Q Eye Module as a comprehensive, procedure- and disease-specific patient-reported outcome instrument.

ELIGIBILITY:
Inclusion criteria

* Women and men between 18-99 years
* With bilateral dermatochalasis and resulting visual field restriction
* Willingness and ability to comply with regular visits
* Signed informed consent form

Exclusion criteria

* Any disease affecting wound closure/healing such as diabetes, connective tissue disease or non-medically induced bleeding disorders, known autoimmune disease, known tendency for hypertrophic scars or keloids;
* Untreated hypertension or metabolic syndrome,
* Smoker
* Asymmetric brow ptosis,
* Previous surgery on the eye lids
* Sequelae after facial nerve palsy
* Allergy or adverse reaction to any substance or material used.
* Active or chronic eyelid inflammation

Pregnant or breast-feeding women:

Women of childbearing potential (18-50) are not excluded form this study. Breastfeeding or pregnant women are however excluded, as bilateral upper eye lid blepharoplasty can be easily postponed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ninety patients will be enrolled in the study. Eligibility will be assessed at the first visit based on inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Overall patient satisfaction | 3 months
  Questionaire: FACE-Q eye module

SECONDARY OUTCOMES:
FACE-Q eye module: individual questions | 3 months
  Questionaire: FACE-Q eye module

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No